CLINICAL TRIAL: NCT03470233
Title: Post-marketing Registry to Assess Usage Information, Safety and Effectiveness of Deltyba® Tablets in Korean Patients With Pulmonary Multi-drug Resistant Tuberculosis (MDR-TB)
Brief Title: Post Marketing Registry to Assess Usage, Safety and Effectiveness of Deltyba Tablets in Korean Patients With MDR-TB
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 242-402-00005
Record Dates: First submitted 2018-02-06; First posted 2018-03-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Multi-drug Resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Deltyba Registry aims to collect the usage information of Deltyba which could be a factor of developing resistance in actual clinical settings.

DETAILED DESCRIPTION:
To collect the usage information of Deltyba in actual clinical settings for the management of resistance to Deltyba

ELIGIBILITY:
Inclusion Criteria

1. Patients who are prescribed Deltyba® per prescribing information (PI) for the purpose of treatment can be included in the registry.

Exclusion Criteria

1. Patients with known hypersensitivity to Delamanid or any excipients of Deltyba®
2. Patients whose serum albumin < 2.8 g/dL
3. Patients taking medicinal products that are strong inducers of CYP3A (e.g. carbamazepine).
4. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption should not take this medicinal product.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are prescribed Deltyba® per prescribing information (PI) for the purpose of treatment can be included.
  The expected number of patients during the enrollment period is 248 patients based on the number of patients who might be taking Deltyba, which was estimated considering annual mean change rate from 2009 to 2014 and the rate of patients who had no resistance to pulmonary MDR-TB therapies2, 3.
  Therefore, the target number of subjects is about 150, which is 60 % of the number of patients who are expected to take Deltyba during the registration period (n=248).
  The number of subjects may vary from one investigator to another.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Dose of Deltyba | for 24 weeks
  Mean values
Administration duration of Deltyba | for 24 weeks
  Mean values
Compliance of Deltyba | for 24 weeks
  percentages (%) of subjects who take Deltyba in excess of 80% compared with the amount of Deltyba prescribed by investigators

SECONDARY OUTCOMES:
Incidences of AEs | at least 1 month after the final administration or premature discontinuation
  Numbers (n) of subjects with AEs
Incidences of ADRs | at least 1 month after the final administration or premature discontinuation
  Percentages (%) of subjects with ADRs
Incidences of AEs in special populations | at least 1 month after the final administration or premature discontinuation
  Percentages (%) of subjects with AEs in special populations, such as the elderly, pregnant women, and patients with hepatic or renal disorder
Incidences of ADRs in special populations | at least 1 month after the final administration or premature discontinuation
  Number (n) of subjects with ADRs in special populations, such as the elderly, pregnant women, and patients with hepatic or renal disorder
Observed cases of resistance to Deltyba after completing the administration (Week 24) or premature discontinuation of Deltyba, Observed cases of resistance to Deltyba after 6 months of administration or discontinuation of administration | after completing the administration (Week 24) or premature discontinuation of Deltyba
  Numbers (n) of subjects who developed drug resistance as determined by drug susceptibility testing (DST) to Deltyba in subjects who resulted in positive in sputum test after termination of the administration or were reverter during the course of treatment
Response rate | at 24 week (at the end of Deltyba administration)
  Number (n) of treatment responders (sustained converters plus new converters), Numbers (n) of sustained converters, new converters, non-converters, and reverters

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan